CLINICAL TRIAL: NCT02941562
Title: A Prospective Phase II Randomized Clinical Trial of Preoperative Chemotherapy Combined With Short-course Radiotherapy Versus Conventional Neo-adjuvant Therapy for Locally Advanced Rectal Cancer Implemented by MDT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Long Cui, Chief Director of Colorectal Surgery, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHGC-004
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Cancer, Radiotherapy
Keywords: rectal cancer, radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

ARMS (2):
- Preoperative chemotherapy with short-course radiotherapy (Experimental): Preoperative treatment:4 course of FOLFOX4 therapy combined with short-course radiotherapy
  Interventions: Radiation: Short-course radiotherapy; Drug: FOLFOX4 chemotherapy,preoperative; Procedure: Radical rectal cancer resection; Drug: FOLFOX4 chemotherapy,post-operative
- Preoperative neo-adjuvant therapy (Active Comparator): Preoperative treatment:neo-adjuvant therapy
  Interventions: Radiation: Radiotherapy of neo-adjuvant therapy; Drug: Concurrent chemotherapy of neo-adjuvant therapy; Procedure: Radical rectal cancer resection; Drug: FOLFOX4 chemotherapy,post-operative

INTERVENTIONS:
Radiation: Short-course radiotherapy — Preoperative Radiation doses: 25 Gy in 5 fractions to the pelvis
  Arms: Preoperative chemotherapy with short-course radiotherapy
Drug: FOLFOX4 chemotherapy,preoperative — FOLFOX4 chemotherapy：5-FU 400 mg/m2 i.v. bolus and Leucovorin 200 mg/m2 i.v. followed by 5-FU 600 mg/m2 i.v. 22 h-infusion day 1 + 2, oxaliplatin 85 mg/m2 day 1.
  Repeat every 2 weeks
  Arms: Preoperative chemotherapy with short-course radiotherapy
Radiation: Radiotherapy of neo-adjuvant therapy — Preoperative Radiation doses: 45 Gy in 25 fractions to the pelvis, 5.4 Gy in 3 fractions to the pelvis
  Arms: Preoperative neo-adjuvant therapy
Drug: Concurrent chemotherapy of neo-adjuvant therapy — Capecitabine 825mg/m2 twice daily 5 days/week
  Arms: Preoperative neo-adjuvant therapy
Procedure: Radical rectal cancer resection — Radical rectal cancer resection
Drug: FOLFOX4 chemotherapy,post-operative — FOLFOX4 chemotherapy：5-FU 400 mg/m2 i.v. bolus and Leucovorin 200 mg/m2 i.v. followed by 5-FU 600 mg/m2 i.v. 22 h-infusion day 1 + 2, oxaliplatin 85 mg/m2 day 1.
  Repeat every 2 weeks

SUMMARY:
The study is designed to analyze the pathological tumor response on locally advanced rectal cancer after preoperative treatment with neo-adjuvant therapy regimen or with chemotherapy combined with short-course radiotherapy in a prospective cohort and to correlate this response with patient's outcome

DETAILED DESCRIPTION:
This is a phase II , open label, randomized study in patients with confirmed diagnosis of locally advanced rectal cancer. The study is designed to analyze the pathological tumor response on locally advanced rectal cancer after preoperative treatment with neo-adjuvant therapy regimen or with chemotherapy combined with short-course radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Consent to this study
* 2. Histological or cytological confirmed diagnostic of rectal carcinoma
* 3. Locally advanced rectal cancer without metastasis, confirmed by pelvic MRI (cT3CRM+、cT4NX or cTxN2M0)(cT3CRM+: margin between the deepest point of tumor and rectal adventitia/serosa surface is less than 1 mm measured in pelvic MRI)
* 4.With no presence of anemia (Hb≤60g/l) induced by tumor bleeding or bowel obstruction
* 5.With no presence of other organ metastasis or extra-regional lymph node involvement
* 6.With no history of chemotherapy
* 7.ECOG score is 0 or 1
* 8.Adequate ability of bone marrow, liver and kidney function
* 9.No pregnancy

Exclusion Criteria:

1. Unable to intake oral medicine
2. Arrhythmia need treatment(besides β-blocker or digoxin); Symptomatic coronary artery disease or history of myocardiac infarction within 6 months ；Congestive Heart Failure NYHA II grade or severe
3. HIV infection or Active chronic HBV or HCV
4. Severe clinical infection at active stage
5. Epileptic seizure need treatment
6. History of organ transplantation
7. Renal failure or intaking renal dialysis
8. Clinical hemorrhagic tendency or Disorders of blood coagulation or intaking anticoagulant or thrombolytics
9. Severe unhealed wound or skin ulcer or bone fraction
10. Measurable massive ascites 11 History of other malignant tumor(except cured cervical tumor in site and cured cutaneous basal cell carcinoma) in last 5 years

12.Chronic inflammatory bowel disease， bowel obstruction，hereditary fructose intolerance 13.Medicine abuse；medical，psychologic or social conditions might disturb patients or results 14.Known or suspected allergy to any drugs in this study 15.Any situation or status that might endanger patient's safety or compliance 16.Pregnant woman or suckling period woman; Fertility without taking sufficient contraception 17.History of pelvic radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Response | Surgery
  Treatment effects of interventions. The tumor response should be graded on a scale of 0 (complete response- no viable cancer cells observed) to 3 (poor response - minimal or no tumor kill; extensive residual cancer)

SECONDARY OUTCOMES:
3-year Disease-Free Survival | 3 years
  time from radical resection to recurrence or end of follow-up
3-year Overall Survival | 3 year
  time from radical resection to cancer caused death or end of follow-up